CLINICAL TRIAL: NCT07336927
Title: Efficacy and Safety of Endovascular Therapy With Intra-Arterial Thrombolysis for Medium Vessel Occlusion Stroke--the IAT-MeVO Trial
Brief Title: IAT-MeVO Trial Domain Within the ACT-GLOBAL Adaptive Platform Trial
Acronym: IAT-MeVO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bo Wu (Other)
Collaborators: West China Hospital (Other); Mianyang Central Hospital (Other); Chengdu First People's Hospital (Other); Sichuan Provincial People's Hospital (Other); Deyang People's Hospital (Other); Suining Central Hospital (Other); The Second People's Hospital of Chengdu (Other)
Responsible Party: Sponsor-Investigator, Bo Wu, Chief Physician/Clinical Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025(No.2695)
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke Due to Medium-vessel-occlusion
Keywords: Acute Ischemic Stroke; Medium vessel occlusion; Intra-arterial thrombolysis; Endovascular therapy; Randomized clinical trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open-label trial; only the outcome assessors and partial data analysts will be masked to treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular Treatment Group (Experimental): Recieving intra-arterial thrombolysis-based EVT after randomization.
  Interventions: Procedure: Endovascular Treatment
- Best Medical Management Group (No Intervention): Upon enrollment, patients will receive best medical management alone.

INTERVENTIONS:
Procedure: Endovascular Treatment — Patients will receive IAT-based EVT in addition to medical treatment. IAT with TNK will be performed first. If adequate dosing fails to achieve reperfusion, the surgical team may evaluate the need for aspiration or stent retriever thrombectomy. For second-order branches (M2/A1/P1 segments), the number of retrieval attempts must not exceed three; for third-order branches (M3/A2/P2 and beyond), no more than two attempts are allowed.
  *Arterial thrombolysis protocol: Dose: 0.125 mg/kg body weight, maximum 12.5 mg
  *No restrictions will be placed on the choice of aspiration catheters or stent retrievers used in this study.
  Arms: Endovascular Treatment Group

SUMMARY:
IAT-MeVO is an international, multicenter, prospective, randomised, open-label, blinded end-point assessed (PROBE) trial, to evaluate the efficacy and safety of endovascular therapy (EVT) [intra-arterial thrombolysis (IAT)-based] versus best medical management (BMT) in patients with acute ischemic stroke (AIS) due to medium vessel occlusion (MeVO) who are ineligible for intravenous thrombolysis (IV) within 24 h of onset.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 y;
2. Diagnosed as acute ischemic stroke;
3. Isolated medium distal vessel occlusion (i.e. an occlusion of the M2, the M3/M4 segment of the MCA, the A1/ A2/A3 segment of the ACA or the P1/P2/P3 segment of the PCA) confirmed by CT or MR Angiography;
4. Time from onset (or last-seen-well) to randomization < 24h;
5. Has not received intravenous thrombolysis and is considered unsuitable for it based on the treating clinician's assessment.
6. NIHSS ≥ 5, or NIHSS ≤ 4 with disabling deficit (e.g. severe aphasia, hemianopia, hemiplegia/loss of function in one side) or fluctuating symptoms at the time of randomization;
7. For patients within 6 h of onset: No visually apparent hypodensity is observed on non-contrast CT compared with the contralateral white matter, or no hyperintensity is seen on fluid-attenuated inversion recovery (FLAIR) imaging; For patients presenting 6-24 h after onset: A perfusion imaging-based ischemic core mismatch ratio >1.2 and an infarct core volume <50 mL are required;
8. Pre-stroke mRS ≤ 1；
9. Patient/Legally Authorized Representative has signed the Informed Consent form.

Exclusion Criteria:

1. Any evidence of intracranial hemorrhage on qualifying imaging;
2. Concurrent multiple (≥2) intracranial arterial occlusions;
3. Suspected cerebral vasculitis, septic embolism, or infective endocarditis as the cause of vessel occlusion;
4. Suspected arterial dissection;
5. Clinical assessment of conditions unsuitable for interventional therapy (e.g., severe contrast agent allergy or absolute contraindications to iodine contrast agent; severe renal insufficiency, glomerular filtration rate < 30ml/min or serum creatinine > 220μmol/L (2.5 mg/dl));
6. Unsuitable for arterial thrombolytic therapy (e.g., known history of hereditary or acquired hemorrhagic disease and/or platelet count <50×109/L; abnormal coagulation function (INR>1.7); oral anticoagulants were taken within 24 - 48 hours before onset within APTT > 3 times normal; recent medical history or clinical manifestations of brain tumors other than meningiomas);
7. Any terminal disease with life expectancy <1 year;
8. Pregnancy or lactation;
9. Concurrent participation in another investigational drug or device study that could interfere with the present trial;
10. Other circumstances that participation is not deemed appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Excellent functional outcome | 90 days
  The proportion of patients with an modified Rankin Scale (mRS) score of 0-1. The mRS is a clinician-reported measure of global disability widely used to assess outcomes in patients with stroke and other neurological disorders. It ranges from 0 (no symptoms) to 6 (death).

SECONDARY OUTCOMES:
Good functional outcome | 90 days
  The proportion of patients with an modified Rankin Scale (mRS) score of 0-2. The mRS is a clinician-reported measure of global disability widely used to assess outcomes in patients with stroke and other neurological disorders. It ranges from 0 (no symptoms) to 6 (death).
Distribution of functional outcome | 90 days
  The modified Rankin Scale (mRS) score at 90 days and the utility weighted mRS. The mRS is a clinician-reported measure of global disability widely used to assess outcomes in patients with stroke and other neurological disorders. It ranges from 0 (no symptoms) to 6 (death).
Health-related quality of life (HRQoL) | 90 days
  Quality of life measured using EQ-5D-5L.The EuroQol 5-Dimension 5-Level instrument (EQ-5D-5L) is a generic, preference-based measure of health-related quality of life. It generates two primary scores: 1) a utility index score (typically ranging from -0.573 to 1.00, depending on the value set, where 1 represents 'full health'), and 2) a self-rated Visual Analog Scale (EQ-VAS) score (ranging from 0 to 100). For both scores, a higher value indicates a better health outcome.
Neurological status | 72±12 hours
  Neurological status measured by National Institutes of Health Stroke Scale (NIHSS) score. The National Institutes of Health Stroke Scale (NIHSS) is a standardized 15-item neurologic examination tool used to quantify the severity of acute cerebral infarction. Scores range from 0 to 42, with higher scores indicating more severe neurological deficit.
Early neurological improvement | 72±12 hours
  Achieving an NIHSS score of 0-1 or a decrease of ≥4 points from the baseline NIHSS score. The National Institutes of Health Stroke Scale (NIHSS) is a standardized 15-item neurologic examination tool used to quantify the severity of acute cerebral infarction. Scores range from 0 to 42, with higher scores indicating more severe neurological deficit.
Final infarct volume | 24-72 hours
  Final infarct size based on CT or MRI
Symptomatic intracranial hemorrhage (sICH) | 7 days
  sICH defined by SIST-MOST criteria
Any intracranial hemorrhage | 7 days
  Any intracranial hemorrhage was a key safety outcome, encompassing any acute bleeding within the cranial cavity. All suspected events were confirmed by follow-up CT or MRI scans.
Malignant cerebral edema | 7 days
  The incidence of malignant edema, adjudicated by the central imaging core lab according to follow-up imaging and medical history
All-cause mortality | 7 days
  Death
All-cause mortality | 90 days
  Death
EVT-related adverse events | 4 days
  adverse events post-EVT

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
This study will include individual information from multicenter and multination. To protect the participants' privacy and follow the guidelines of other center or nations' ethical committee, we don't provide or share IPD with other reasearchers.